CLINICAL TRIAL: NCT06422026
Title: A 24 Week, Randomized, Double Blind, Placebo Controlled Clinical Trial for the Evaluation of the Efficacy and Safety of APCP on Hair Health
Brief Title: Evaluated the Efficacy and Safety of APCP on Hair Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AP-PV-2022-02
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Hair Damage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- APCP I (Active Comparator)
  Interventions: Dietary Supplement: APCP I
- APCP II (Active Comparator)
  Interventions: Dietary Supplement: APCP II
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: APCP I — Each subject takes one active bottle per day for 24 weeks. Each bottle contains APCP 3 g.
  Arms: APCP I
Dietary Supplement: APCP II — Each subject takes one active bottle per day for 24 weeks. Each bottle contains APCP 4 g.
  Arms: APCP II
Dietary Supplement: Placebo — Each subject takes one active bottle per day for 24 weeks.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy and safety of APCP in promoting hair health in adult with mild to moderate hair damage, compared to a placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Glossy scores according to the visual evaluation classification method correspond to 1 point or more and 3 points or less and a total hair damage score of less than 18 points evaluated according to exposure to risk factors
* A person capable of maintaining the same hair shape and color during this human body application test
* A person who has agreed to participate in this human application test before the start of the human application test and filled out the Informed Consent Form

Exclusion Criteria:

* A person currently being treated for infectious diseases and malignant tumors, including severe cardiovascular system, immune system, respiratory system, hepatometer, kidney and urology system, nervous system, musculoskeletal system, psychosis, skin, etc
* As of Visit 1, those who currently have dull dermatitis, scalp psoriasis, and scalp infection
* A person who plans to manage and operate hair supplies, hair products during this human body application test
* A person who has taken oral Dutasteride or Finasteride within 6 months of visit 1
* A person who has applied topical hair growth agents, wool, and hair growth agents for the last 1 month (30 days) or more as of Visit 1
* Those who have been administered systemic steroids, cell death agents, vasodilators, antihypertensive agents, antiepileptic agents, beta receptor blockers, bronchodilators, diuretics, Cimetidine, Diazoxide, Cyclosporine, and Ketoconazole for the last 1 month or more (30 days)
* A person who has applied topical steroids to the scalp for the last 1 month (30 days) or more as of Visit 1
* A person who has participated in other interventional clinical trials (including human application tests) within one month (30 days) of visit 1 or plans to participate in other interventional clinical trials (including human application tests) after the start of this human application test
* A person who is pregnant or who has a plan to become pregnant during the nursing mother or during this human body application test
* A person who is sensitive to or allergic to food ingredients for this human body application test
* A person who is deemed inappropriate by the tester for other reasons

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hair tensile strength | Baseline, 24 week
  Hair tensile strength measured by UTM(Universal Testing Machine) etc.

SECONDARY OUTCOMES:
Change from baseline in hair gloss | Baseline, 24 week
  Hair gloss measured by Glossymeter etc.
Change from baseline in hair density | Baseline, 24 week
  Hair density measured by Folliscope
Change from baseline in hair volume | Baseline, 24 week
  Hair volume measured by I Max-plus
Change from baseline in satisfaction survey | Baseline, 24 week
  Satisfaction surveys are evaluated on a 10-point scale. Survey items are evaluated on a scale from '0 - Not at all' to '10 - Very much so' (although scoring may be reversed depending on the question).
Change from baseline in scalp moisture | Baseline, 24 week
  scalp moisture measured by DermaLab Hydration Pin Probe
Change from baseline in scalp percutaneous moisture loss | Baseline, 24 week
  scalp percutaneous moisture loss measured by Tewameter TM Nano

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No